CLINICAL TRIAL: NCT01079494
Title: Clinical Pharmacists Role in the Management of Hypertension in Jordan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Jordan Hospital (Other)
Responsible Party: Eman Hammad, faculty of pharmacy / University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JU8071383
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2009-03

CONDITIONS: Hypertension
Keywords: Uncontrolled blood pressure
MeSH Terms: conditions — Hypertension | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Active Comparator): physician-pharmacist teamwork
  Interventions: Other: pharmaceutical care services
- control (No Intervention): physician only team

INTERVENTIONS:
Other: pharmaceutical care services — Patients treatment related problems and therapeutic needs or complains identified by clinical pharmacist and managed collaboratively by both pharmacist and the physician.
  Arms: intervention group

SUMMARY:
Background: studies have demonstrated the crucial role of clinical pharmacists as integrated part of heath care team. Not only in Jordan but also in the Middle East region, clinical pharmacy practice is not well established. This current study is the first to evaluate physicians - pharmacists' collaborative approach to uncontrolled blood pressure in Jordan and the Middle East.

DETAILED DESCRIPTION:
Objective: this study aimed to evaluate clinical pharmacists' role in the management of uncontrolled hypertensive patients in Jordan. Design: single blinded randomized controlled clinical trial. Patients: 253 patients with uncontrolled hypertension specified as higher blood pressure readings than the recommended goals by the seventh report of the Joint National Committee on prevention, detection, evaluation, and treatment of high blood pressure (JNC VII) at the time of enrollment.

Interventions: patients were randomly allocated to an intervention or control group: 130 and 123 patients, respectively. Patients in both arms were followed up for 6 months. In the intervention group, patients were managed by physician-clinical pharmacist team. In the control group, patients were managed by physician(s) only and were not provided pharmaceutical care services.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled BP, receiving 0-3 antihypertensive drugs with no change in the regimen or dose within the past 3 month.

Exclusion Criteria:

* Patients with hypertensive urgency or emergency with BP more than (180/110).
* Patients with recent stroke or myocardial infraction (within past 6 months).
* Patients with Class III or IV Chronic heart Failure (CHF).
* Patients with Unstable angina.
* Patients with Serious renal or hepatic disease.
* Pregnant patients.
* Patients with Dementia or cognitive impairment.
* If the patient is unable to provide informed written consent.

Ages: 21 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
percentage of patients who achieved blood pressure goals specified by the JNC VII at each group | 6 month
  defined a goal to be achieved if the systolic blood pressure fell below 140 mm Hg and the diastolic blood pressure fell below 90 mm Hg. Or systolic blood pressure fell below 130 mm Hg and the diastolic blood pressure fell below 80 mm Hg if patient was diabetic.

SECONDARY OUTCOMES:
mean reductions in both systolic and diastolic blood pressure readings | 6 months
  mean reductions in systolic blood pressure (Systolic blood pressure at enrollment - Systolic blood pressure last follow up visit) and diastolic BP (Diastolic blood pressure at enrollment - Diastolic blood pressure last follow up visit) for both study groups

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hammad, MSc, Principal Investigator — University of Jordan/ Faculty of Pharmacy; Abla Al bsoul, PhD, Study Director — University of Jordan/ Faculty of Pharmacy
Locations (1):
- family medicine clinic JUH, Amman, Jordan